CLINICAL TRIAL: NCT00284648
Title: Operative Versus Non-operative Treatment of Achilles Tendon Rupture: A Multicentre, Prospective Randomized Study.
Brief Title: Operative Versus Non-operative Treatment of Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fowler Kennedy Sport Medicine Clinic (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Sharon Griffin, Research Coordinator, Fowler Kennedy Sport Medicine Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 99-36
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon; Rupture; Non-operative; Operative
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Surgical repair Achilles tendon rupture
Procedure: Non-surgical repair Achilles tendon rupture

SUMMARY:
This study is intended to determine whether the optimal treatment of acute Achilles tendon ruptures is surgical repair or functional bracing.

Our hypotheses are surgical repair will: 1) Result in a clinically relevant decrease in re-rupture rate and 2) Result in a clinically relevant improvement in disease specific quality of life and 3) A clinically relevant improvement in functional outcome measures

DETAILED DESCRIPTION:
Methodology This study is a multi-centre prospective randomized controlled clinical trial. This study will be conducted at five tertiary care centres by orthopaedic surgeons with an interest in soft tissue trauma. All subjects will be recruited over a one year period. Subjects who meet the following inclusion and exclusion criteria and who consent to involvement in the study will be randomized to either operative or non-operative arms of the study. All patients who enter the study will receive a pre-treatment ultrasound to document that the tear is complete and to document the location of the tear. Prior to obtaining consent for the study the risks and benefits of each treatment option will be clearly explained along with the current state of knowledge concerning treatment of Achilles tendon ruptures. It will be explained to each study participant that involvement in the study is voluntary and that they are free to discontinue their involvement at any point in their treatment .

Inclusion Criteria

* Complete Achilles Tendon Rupture
* Less than 7 days from date of injury
* Age 18-70 years of age
* Ability to follow rehab protocol

Exclusion Criteria

* Inability to Speak English
* Significant ipsilateral injury
* Open injury to Achilles tendon
* Neurological disease (ie stroke, cerebral palsy)
* Collagen Disease (ie Ehlers Danlos disease)
* Pregnancy
* Fluoroquinolone associated rupture (rupture within 2 weeks of taking medication)
* Unfit for surgery
* Diabetes
* Peripheral Vascular disease
* Avulsion of Achilles tendon from calcaneus

Surgical Repair If randomized to the operative group, all patients will be evaluated and informed consent obtained. Surgery will performed as outpatient day surgery. Prophylactic antibiotics will be given one hour prior to the procedure. All patients will receive general anaesthesia and endotracheal intubation. The patient will be positioned prone on bolsters on the operative table. A tourniquet will be applied to the thigh of the affected extremity and inflated to 300 mmHg at the start of the case.

The affected limb will be prepared and draped in the standard fashion. A medial to lateral curvilinear incision will be utilzed. The posterior aspect of the tendon and tendon sheath will then be exposed. Evacuation of the overlying clot will then expose the ruptured tendon. Two ethibond sutures will be placed in each end of the torn tendon (total of four sutures). Two ethibond sutures will be placed in a modified Bunnel stitch fashion entering at the tear site, first going proximally towards normal tendon and then distally towards the calcaneus. With the foot in neutral alignment the sutures will be tied proximally and distally in normal tendon away from the tear site. A 2-0 vicryl suture will then be place at the site of the repair in a running fashion to augment the repair. The wound will be irrigated and the tendon sheath will be closed with a running 2-0 running vicryl stitch. The skin will be closed with interrupted 3-0 nylon suture and a sterile dressing and tubigrip applied.

In the recovery room the patient will be fitted with a plaster backslab in gravity plantar flexion (approx. 20 degrees).

Postoperative Protocol Patients will be instructed to be non-weight bearing on their injured side with crutch assistance until seen in the outpatient clinic in 7-10 days. Patients will then be fitted for and Air Cast Boot splint. Patients will then be instructed to be weight bearing as tolerated on their injured side with crutch assistance for a period of six weeks.

Patients will be allowed active plantar flexion and dorsiflexion up to neutral with physiotherapy supervision. The Air Cast Boot will be removed for therapy but should be worn otherwise for protection. At six weeks patients will have their splints removed and be allowed to weight bear as tolerated. At the six week interval patients will also begin to perform dorsiflexion stretching exercises and will begin graduated resistance exercises. Follow up appointments will be 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years following surgery.

Functional Bracing Treatment If randomized to the functional bracing group, subjects will have an Air Cast Boot splint applied with a 2cm felt heel lift. Ath two weeks the heel lift will be removed. As with the operative group patients will be weight bearing as tolerated on their injured side with crutch assistance for six weeks. Similarly, subjects will be allowed to remove the Air Cast Boot and perform active plantar flexion and dorsiflexion up to neutral with physiotherapy supervision. At six weeks the patients will have their Cast Boots removed and dorsiflexion stretching exercises will be begun. A gentle resistance program will also begin at six weeks along with dorsiflexion stretching exercises. Follow up appointments will be 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years following the initial injury.

Re-rupture Rate and Complications The primary outcome measure will be re-rupture rate. This will be determined at follow-up intervals of: 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years

Re-rupture rates between the operative and non-operative groups will be calculated and statistically analysed using a student's t test. P values of less than 0.05 will be considered significant. Any clinical suspicion of a re-rupture will require an ultrasound for confirmation. Re-ruptures will be treated surgically. At the above listed follow-up intervals other complications will also be recorded including:

Minor complications

* superficial infection
* wound hematoma
* delayed wound healing
* scar adhesion
* sensory disturbances
* suture granuloma

Major Complications

* re-rupture
* equinus postioning of foot
* extreme lengthening of tendon
* deep infection
* chronic fistula
* necrosis of skin
* deep vein thrombosis
* embolism
* death

Range of Motion, Strength and Calf Circumference Range of motion and calf circumference will be documented at 6 weeks, 3 months, 6 months, 1 year and 2 years. Active range of motion only will be recorded to avoid healing setbacks. Calf circumference will be recorded and compared to the unaffected extremity.

Strength Testing Strength testing will be performed on all study participants. This will be done at follow-up visits at 6 months, 1 year and 2 years. These measurements will include peak torque and total work. A cybex dynamometer will be used to test isokinetic concentric plantar and dorsiflexion strength at 30, 90 and 240 degrees per second. All values will be compared to the opposite unaffected side. Scores will then be transformed into a percentage of the unaffected side and points awarded appropriately as per the outcome measure designed by Leppilahti et al.

Disease Specific Quality of Life In the debate surrounding the most effective management of Achilles tendon ruptures, surgeons have argued about which individual factor signifies success. Many authors have suggested that re-rupture rate should be considered the measure of successful treatment, while others suggest minor complications or return to sport may also warrant consideration.

This study will utilize a previously published outcome scoring system that attempts to evaluate important factors in the recovery from this injury. This measurement tool published by Leppilahti et al utilizes a combination of factors including pain, stiffness and footwear restrictions as well as objective strength values, to arrive at an overall score. Statistical analysis using a students t test will be applied to the outcome score means of the operative and non-operative groups. P values of less than 0.05 will be considered significant. The application of this scoring system to a prospective randomized trial comparing operative and non-operative treatment of this condition will hopefully shed some much needed light on this therapeutic dilemma.

ELIGIBILITY:
Inclusion Criteria:

* Complete Achilles Tendon Rupture Less than 7 days from date of injury Age 18-70 years of age Ability to follow rehab protocol

Exclusion Criteria:

Inability to Speak English Significant ipsilateral injury Open injury to Achilles tendon Neurological disease (ie stroke, cerebral palsy) Collagen Disease (ie Ehlers Danlos disease) Pregnancy Fluoroquinolone associated rupture (rupture within 2 weeks of taking medication) Unfit for surgery Diabetes Peripheral Vascular disease Avulsion of Achilles tendon from calcaneus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Re-rupture rate

SECONDARY OUTCOMES:
Minor complications
Major Complications
Range of Motion, Strength and Calf Circumference
Strength Testing
Disease Specific Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Willits, MD, Principal Investigator — The University of Western Ontario
Locations (1):
- Fowler Kennedy Sport Medicine Clinic, University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Willits K, Amendola A, Bryant D, Mohtadi NG, Giffin JR, Fowler P, Kean CO, Kirkley A. Operative versus nonoperative treatment of acute Achilles tendon ruptures: a multicenter randomized trial using accelerated functional rehabilitation. J Bone Joint Surg Am. 2010 Dec 1;92(17):2767-75. doi: 10.2106/JBJS.I.01401. Epub 2010 Oct 29. PMID 21037028